CLINICAL TRIAL: NCT03657238
Title: A Phase 1, Randomised, Double-blind, Single-centre, Placebo-controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single S.C. Doses of RD01 (Pegerythropoietin) in Healthy Chinese Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of RD01 (Pegerythropoietin) in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shengzhen Sciprogen Bio-pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3SBio-RD01-101a
Record Dates: First submitted 2018-08-24; First posted 2018-09-05 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Doses were escalated from 0.2μg/kg up to 4.8μg/kg
  Interventions: Drug: RD01
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RD01 — single S.C. dose of RD01 for subjects in test group
  Arms: Experimental
Drug: Placebo — single S.C. dose of placebo for subjects in placebo group
  Arms: Placebo

SUMMARY:
A first-time in human study to investigate the safety, tolerability and pharmacokinetics of RD01 in healthy Chinese subjects

DETAILED DESCRIPTION:
A Phase 1, Randomised, Double-blind, Single-centre, Placebo-controlled, Dose-Escalation study to evaluate the Safety, Tolerability and Pharmacokinetics of single S.C. doses of RD01 (Pegerythropoietin) in Healthy Chinese Subjects. Doses were escalated from 0.2μg/kg up to 4.8μg/kg with 12 subjects (randomized to 5:1 for test or placebo) in every cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~60, both male and female
* Healthy adults without obvious organic diseases and nervous/mental diseases
* BMI 19~26 kg/m2, inclusive
* Subject is willing and able to provide written informed consent, and would complete the whole study procedures
* Serum ferritin level is within the reference range at screening within 4 weeks before enrollment
* Should be fully recovered, when has received surgical treatment

Exclusion Criteria:

* Has allergy history or past drug allergy history, or allergy history to polyethylene glycol
* Has taken any drug within 5 half-time or 4 weeks before enrollment
* Has taken any drug known to harm organ within 12 weeks before enrollment
* Participated in other clinical trials within 12 weeks before enrollment
* Donated blood or received blood transfusion, or received therapy of recombinant erythrocytogenetic stimulating protein or rHuEPO within 12 weeks before enrollment
* Female subject receives therapy of hormone after menopause
* Subject with clinically significant abnormal of lab tests determined by the investigator (subjects with Hb or Rtc level outrange the up-limit of reference were suggested to be excluded)
* Subject with HBsAg, HBeAg, HCV-Ab, HIV-Ab or Treponema pallidum antibody positive
* Clinically diagnosed as vitamin B12 or folic acid deficiency
* Previous history of coronary heart disease or congestive heart failure, or ECG shows clinical significance of abnormalities
* With history of malignant tumors or suspicious
* Subject with active infection
* History of autoimmune disease, or being treated with immunosuppressive agents
* With severe, progressive or uncontrolled diseases of liver, kidney, blood, gastrointestinal tract, endocrine, heart, lung, nerves or brain
* Pregnant or lactating women, or subject planning to has descendants during trial or within 12 weeks after dosing
* Drug abusers, drug addicts, or smokers (5 or more cigarettes per day), alcoholics (14 or more units per week, 1 unit = 360 mL of beer or 150 mL of wine or 45 mL of alcohol 40% or more)
* Other factors that might influence the attendance determined by investigators, including poor compliance (long-term travel, planned relocation, mental illness, lack of motivation, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
incidence of Adverse Events | up to 35 days
  incidence of adverse events using the NCI Common Terminology Criteria for Adverse Events version 4.0.

SECONDARY OUTCOMES:
maximum concentration （Cmax） | for 35days
  Plasma RD01 concentration will be quantified for each arm to determine Cmax, defined as the maximum observed concentration of RD01 in plasma.
time to reach Cmax （Tmax） | for 35days
  Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them
terminal elimination half life（t½） | for 35days
  It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase.
the changes of hemoglobin (g/L) after treatment | for 35days
  The hemoglobin of participants the was measured before and after the treatment
the changes of reticulocyte (10^9/L) after treatment | for 35days
  The reticulocyte of participants the was measured before and after the treatment
the changes ofHematocrit（%） after treatment | for 35days
  The Hematocrit of participants the was measured before and after the treatment
the changes of erythrocyte（10^12/L） after treatment | for 35days
  The erythrocyte of participants the was measured before and after the treatment

OTHER OUTCOMES:
Anti-drug antibody endpoint | up to 35 days
  Blood level for anti-EPO and anti-RD01 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Hu C, Sun W, Wu Y, Huang J, Zhang X, Zhang L. A Phase I Dose-Escalation Study of The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Polyethylene Glycol-Erythropoietin (PEG-EPO) in Healthy Subjects. Clin Ther. 2024 Aug;46(8):636-643. doi: 10.1016/j.clinthera.2024.06.018. Epub 2024 Aug 8. PMID 39117488